CLINICAL TRIAL: NCT05366738
Title: A Phase 1, Open-label, Randomized, Single-dose, Crossover Study to Determine the Bioavailability of Vonoprazan Sprinkle Capsules on Pudding or on Applesauce Relative to a Vonoprazan Tablet in Healthy Participants
Brief Title: A Study to Determine the Bioavailability of Vonoprazan Sprinkle Capsules on Pudding or on Applesauce Relative to a Vonoprazan Tablet in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Phathom Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: VPED-101
Record Dates: First submitted 2022-05-04; First posted 2022-05-09 (Actual); Results first posted 2024-03-29 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2023-09

CONDITIONS: Healthy Volunteers
Keywords: Vonoprazan; Gastroesophageal Reflux; Erosive Esophagitis
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Treatment Sequence 1 (Experimental): Participants assigned to Treatment Sequence 1 will receive vonoprazan 20 mg as a sprinkle capsule on 1 tablespoon of pudding on Day 1 of Treatment Period 1, vonoprazan 20 mg as a sprinkle capsule on 1 tablespoon of applesauce on Day 1 of Treatment Period 2, and vonoprazan 20 mg as a tablet on Day 1 of Treatment Period 3.
  Interventions: Drug: Vonoprazan
- Treatment Sequence 2 (Experimental): Participants assigned to Treatment Sequence 2 will receive vonoprazan 20 mg as a tablet on Day 1 of Treatment Period 1, vonoprazan 20 mg as a sprinkle capsule on 1 tablespoon of pudding on Day 1 of Treatment Period 2, and vonoprazan 20 mg as a sprinkle capsule on 1 tablespoon of applesauce on Day 1 of Treatment Period 3.
  Interventions: Drug: Vonoprazan
- Treatment Sequence 3 (Experimental): Participants assigned to Treatment Sequence 3 will receive vonoprazan 20 mg as a sprinkle capsule on 1 tablespoon of applesauce on Day 1 of Treatment Period 1, vonoprazan 20 mg as a tablet on Day 1 of Treatment Period 2, and vonoprazan 20 mg as a sprinkle capsule on 1 tablespoon of pudding on Day 1 of Treatment Period 3.
  Interventions: Drug: Vonoprazan

INTERVENTIONS:
Drug: Vonoprazan — Orally via tablet
Drug: Vonoprazan — Orally via sprinkle pellets

SUMMARY:
The primary objective of this study is to assess the bioavailability (BA) of a single oral dose of vonoprazan 20 mg sprinkle capsule, either sprinkled on pudding or on applesauce, relative to a vonoprazan 20 mg tablet in healthy participants.

DETAILED DESCRIPTION:
This clinical trial information was submitted voluntarily under the applicable law and, therefore, certain submission deadlines may not apply. (That is, clinical trial information for this applicable clinical trial was submitted under section 402(j)(4)(A) of the Public Health Service Act and 42 CFR 11.60 and is not subject to the deadlines established by sections 402(j)(2) and (3) of the Public Health Service Act or 42 CFR 11.24 and 11.44.).

ELIGIBILITY:
Inclusion Criteria:

* The participant is male or female 18 to 55 years of age, inclusive, at Screening.
* The participant has a body mass index 18 to 32 kg/m^2, inclusive, at Screening.
* The participant is considered by the investigator to be in good general health as determined by medical history, clinical laboratory test results, vital sign measurements, 12-lead ECG results, and physical examination findings at Screening.
* Male and female participants of reproductive potential must use an acceptable method of birth control (i.e., diaphragm with spermicide, intrauterine device, condom with foam or vaginal spermicide, oral contraceptives, or abstinence) from the signing of informed consent until 4 weeks after the last dose of study drug or be surgically sterile (i.e., vasectomy, hysterectomy, bilateral tubal ligation or bilateral oophorectomy) or postmenopausal (defined as amenorrhea for 12 consecutive months and documented plasma follicle stimulating hormone [FSH] level >40 international unit (IU)/mL during Screening).
* Female participants must have a negative pregnancy test at Screening and upon Check-in.
* The participant agrees to comply with all protocol requirements.
* The participant is able to provide written informed consent.

Exclusion Criteria:

* The participant has a positive test result for hepatitis B surface antigen, hepatitis C virus antibody, or human immunodeficiency virus types 1 or 2 antibodies at Screening.
* The participant has a positive test result for the presence of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) at Screening or Check-in.
* The participant has a history of a clinically significant neurological, cardiovascular, pulmonary, hepatic, renal, metabolic, gastrointestinal, or endocrine disease or other abnormality that may impact the ability of the participant to participate.
* The participant has current or recent (within 6 months) gastrointestinal conditions that would be expected to influence the absorption of drugs (e.g., history of malabsorption, esophageal reflux, peptic ulcer disease, erosive esophagitis [EE]), frequent (more than once per week) occurrence of heartburn, or any surgical intervention.
* The participant has any other clinically significant findings on physical examination, clinical laboratory abnormalities, and/or ECG results that preclude his/her participation in the study, as deemed by the investigator.
* The participant has used any prescription (excluding hormonal birth control) and/or over-the-counter medications (including CYP3A4 inducers) except acetaminophen (up to 2 g per day), including herbal or nutritional supplements, within 14 days before the first dose of study drug, and/or is expected to require any such medication during the course of the study until end of treatment period phase (ET) or end of study (EOS).
* The participant has consumed grapefruit and/or grapefruit juice, Seville orange or Seville orange-containing products (eg, marmalade), or other food products that may be CYP3A4 inhibitors (eg, vegetables from the mustard green family [kale, broccoli, watercress, collard greens, kohlrabi, Brussels sprouts, mustard] and charbroiled meats) within 7 days (or 5 half-lives) before the first dose of study drug and/or is expected to be unable to abstain through the study.
* The participant has consumed caffeine- or xanthine-containing products within 48 hours (or 5 half-lives) before the first dose of study drug and/or is unable to abstain through the study.
* The participant is a smoker and/or has used nicotine or nicotine-containing products (eg, snuff, nicotine patch, nicotine chewing gum, mock cigarettes, or inhalers) within 6 months before the first dose of study drug.
* The participant has a history of alcohol abuse and/or drug addiction within the last year or excessive alcohol consumption (regular alcohol intake >21 units per week for male participants and >14 units of alcohol per week for female participants; 1 unit is equal to approximately 1/2 pint [200 mL] of beer, 1 small glass [100 mL] of wine, or 1 measure [25 mL] of spirits) or use of alcohol 48 hours before the first dose of study drug.
* The participant has a positive test result for drugs of abuse, alcohol, or cotinine (indicating active current smoking) at Screening or Check-in.
* The participant is involved in strenuous activity or contact sports within 24 hours before the first dose of study drug and during the study.
* The participant has donated blood or blood products >450 mL within 30 days before the first dose of study drug.
* The participant has a history of relevant drug and/or food allergies (i.e., allergy to vonoprazan or excipients or any significant food allergy that could preclude a standard diet in the clinical unit).
* The participant has received a study drug in another investigational study within 30 days of dosing.
* Female participants who are pregnant or lactating; intend to become pregnant before, during, or within 4 weeks after participating in this study; or intend to donate ova during this time period.
* The participant is not suitable for entry into the study in the opinion of the investigator.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2022-05-18 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Phathom Pharmaceuticals
Locations (1):
- PPD Development, LP, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 27 participants were randomized in a 1:1:1 ratio to 1 of 3 treatment sequences at 1 site in the United States.
Pre-assignment Details: Screening assessments were conducted within 28 days before randomization.
Groups:
- Vonoprazan 20 mg: Treatment Sequence 1: Participants received vonoprazan 20 mg orally as a sprinkle capsule on 1 tablespoon of pudding on Day 1 of Treatment Period 1, orally as a sprinkle capsule on 1 tablespoon of applesauce on Day 1 of Treatment Period 2, and orally as a tablet on Day 1 of Treatment Period 3. Each treatment period was 3 days, with treatment received on Day 1 of each treatment period. There was a washout interval of a minimum of 7 days between study drug dosing in each period.
- Vonoprazan 20 mg: Treatment Sequence 2: Participants received vonoprazan 20 mg orally as a tablet on Day 1 of Treatment Period 1, orally as a sprinkle capsule on 1 tablespoon of pudding on Day 1 of Treatment Period 2, and orally as a sprinkle capsule on 1 tablespoon of applesauce on Day 1 of Treatment Period 3. Each treatment period was 3 days, with treatment received on Day 1 of each treatment period. There was a washout interval of a minimum of 7 days between study drug dosing in each period.
- Vonoprazan 20 mg: Treatment Sequence 3: Participants received vonoprazan 20 mg orally as a sprinkle capsule on 1 tablespoon of applesauce on Day 1 of Treatment Period 1, orally as a tablet on Day 1 of Treatment Period 2, and orally as a sprinkle capsule on 1 tablespoon of pudding on Day 1 of Treatment Period 3. Each treatment period was 3 days, with treatment received on Day 1 of each treatment period. There was a washout interval of a minimum of 7 days between study drug dosing in each period.
Period: Overall Study
Arm/Group | Vonoprazan 20 mg: Treatment Sequence 1 | Vonoprazan 20 mg: Treatment Sequence 2 | Vonoprazan 20 mg: Treatment Sequence 3
Started | 9 | 9 | 9
Completed Treatment A (Vonoprazan 20 mg Sprinkle Capsule on Pudding) | 9 | 8 | 9
Completed Treatment B (Vonoprazan 20 mg Sprinkle Capsule on Applesauce) | 9 | 8 | 9
Completed Treatment C (Vonoprazan 20 mg Tablet) | 9 | 9 | 9
Completed | 9 | 8 | 9
Not Completed | 0 | 1 | 0
Not completed — Adverse Event | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vonoprazan 20 mg: Treatment Sequence 1 | Vonoprazan 20 mg: Treatment Sequence 2 | Vonoprazan 20 mg: Treatment Sequence 3 | Total
Number analyzed (Participants) | 9 | 9 | 9 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.1 (7.22) | 32.9 (8.51) | 35.8 (9.63) | 34.6 (8.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 4 | 11
  Male | 4 | 7 | 5 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 2 | 3 | 11
  Not Hispanic or Latino | 3 | 7 | 6 | 16
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 2 | 4 | 10
  White | 5 | 6 | 5 | 16
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve From Time 0 to the Last Quantifiable Concentration (AUC0-t) of Vonoprazan
Time Frame: Day 1 of each 3-day Treatment Period: Within 0.25 hours pre-dose and 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 10, 12, 16, 24, 36, and 48 hours post-dose.
Population: Measured in the pharmacokinetic (PK) population, which included all participants who received at least 1 dose of vonoprazan and had sufficient concentration data to support accurate estimation of at least 1 PK parameter. PK data are presented for each treatment received, as pre-specified.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng•h/mL
Groups:
- Treatment A: Vonoprazan 20 mg Sprinkle Capsule on Pudding: Participants received vonoprazan 20 mg orally as a sprinkle capsule on 1 tablespoon of pudding on Day 1 of their assigned Treatment Period. Which treatment the participants received in each Treatment Period was dependent upon which Treatment Sequence they were assigned to at randomization.
- Treatment B: Vonoprazan 20 mg Sprinkle Capsule on Applesauce: Participants received vonoprazan 20 mg orally as a sprinkle capsule on 1 tablespoon of applesauce on Day 1 of their assigned Treatment Period. Which treatment the participants received in each Treatment Period was dependent upon which Treatment Sequence they were assigned to at randomization.
- Treatment C: Vonoprazan 20 mg Tablet: Participants received vonoprazan 20 mg orally as a tablet on Day 1 of their assigned Treatment Period. Which treatment the participants received in each Treatment Period was dependent upon which Treatment Sequence they were assigned to at randomization.
Arm/Group | Treatment A: Vonoprazan 20 mg Sprinkle Capsule on Pudding | Treatment B: Vonoprazan 20 mg Sprinkle Capsule on Applesauce | Treatment C: Vonoprazan 20 mg Tablet
Number analyzed (Participants) | 26 | 26 | 27
ng•h/mL | 228 (44.9) | 216 (46.0) | 219 (47.3)
Statistical Analysis 1: Comparison: Treatment A: Vonoprazan 20 mg Sprinkle Capsule on Pudding vs Treatment C: Vonoprazan 20 mg Tablet; Test type: Equivalence — Bioequivalence was concluded if the 90% confidence interval for the geometric mean ratio between the test treatments (20 mg sprinkle capsule, either sprinkled on pudding or on applesauce) and the reference treatment (20 mg tablet) were wholly contained within 80.00% and 125.00% for the vonoprazan PK parameters; Ratio of Geometric Least Square Means = 103.36, 90% CI 2-sided [97.64 to 109.41]
Statistical Analysis 2: Comparison: Treatment B: Vonoprazan 20 mg Sprinkle Capsule on Applesauce vs Treatment C: Vonoprazan 20 mg Tablet; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of Geometric Least Square Means = 97.83, 90% CI 2-sided [92.42 to 103.56]

2. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve From Time 0 Extrapolated to Infinity (AUC0-inf) of Vonoprazan
Time Frame: as for outcome 1
Population: Measured in the PK population, which included all participants who received at least 1 dose of vonoprazan and had sufficient concentration data to support accurate estimation of at least 1 PK parameter. PK data are presented for each treatment received, as pre-specified.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng•h/mL
Arm/Group | Treatment A: Vonoprazan 20 mg Sprinkle Capsule on Pudding | Treatment B: Vonoprazan 20 mg Sprinkle Capsule on Applesauce | Treatment C: Vonoprazan 20 mg Tablet
Number analyzed (Participants) | 26 | 26 | 27
ng•h/mL | 238 (43.2) | 227 (43.1) | 231 (44.4)
Statistical Analysis 1: Comparison: Treatment A: Vonoprazan 20 mg Sprinkle Capsule on Pudding vs Treatment C: Vonoprazan 20 mg Tablet; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of Geometric Least Square Means = 102.56, 90% CI 2-sided [97.25 to 108.15]
Statistical Analysis 2: Comparison: Treatment B: Vonoprazan 20 mg Sprinkle Capsule on Applesauce vs Treatment C: Vonoprazan 20 mg Tablet; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of Geometric Least Square Means = 97.61, 90% CI 2-sided [92.55 to 102.93]

3. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Vonoprazan
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Treatment A: Vonoprazan 20 mg Sprinkle Capsule on Pudding | Treatment B: Vonoprazan 20 mg Sprinkle Capsule on Applesauce | Treatment C: Vonoprazan 20 mg Tablet
Number analyzed (Participants) | 26 | 26 | 27
ng/mL | 23.1 (44.2) | 22.4 (41.9) | 22.3 (45.3)
Statistical Analysis 1: Comparison: Treatment A: Vonoprazan 20 mg Sprinkle Capsule on Pudding vs Treatment C: Vonoprazan 20 mg Tablet; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of Geometric Least Square Means = 103.96, 90% CI 2-sided [96.49 to 112.00]
Statistical Analysis 2: Comparison: Treatment B: Vonoprazan 20 mg Sprinkle Capsule on Applesauce vs Treatment C: Vonoprazan 20 mg Tablet; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of Geometric Least Square Means = 100.60, 90% CI 2-sided [93.38 to 108.39]

4. Secondary Outcome: Time to Maximum Observed Plasma Concentration (Tmax) of Vonoprazan
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | Treatment A: Vonoprazan 20 mg Sprinkle Capsule on Pudding | Treatment B: Vonoprazan 20 mg Sprinkle Capsule on Applesauce | Treatment C: Vonoprazan 20 mg Tablet
Number analyzed (Participants) | 26 | 26 | 27
hours | 2.00 [1.50 to 6.00] | 2.01 [1.00 to 6.00] | 2.00 [1.50 to 6.02]

5. Secondary Outcome: Terminal Phase Half-life (t1/2) of Vonoprazan
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Treatment A: Vonoprazan 20 mg Sprinkle Capsule on Pudding | Treatment B: Vonoprazan 20 mg Sprinkle Capsule on Applesauce | Treatment C: Vonoprazan 20 mg Tablet
Number analyzed (Participants) | 26 | 26 | 27
hours | 7.50 (19.5) | 7.20 (18.4) | 7.29 (16.0)

6. Secondary Outcome: Apparent Total Body Clearance (CL/F) of Vonoprazan
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: litres/h
Arm/Group | Treatment A: Vonoprazan 20 mg Sprinkle Capsule on Pudding | Treatment B: Vonoprazan 20 mg Sprinkle Capsule on Applesauce | Treatment C: Vonoprazan 20 mg Tablet
Number analyzed (Participants) | 26 | 26 | 27
litres/h | 83.9 (43.2) | 88.1 (43.1) | 86.6 (44.4)

7. Secondary Outcome: Apparent Volume of Distribution (Vz/F) of Vonoprazan
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: litres
Arm/Group | Treatment A: Vonoprazan 20 mg Sprinkle Capsule on Pudding | Treatment B: Vonoprazan 20 mg Sprinkle Capsule on Applesauce | Treatment C: Vonoprazan 20 mg Tablet
Number analyzed (Participants) | 26 | 26 | 27
litres | 908 (37.6) | 915 (33.4) | 911 (38.5)

8. Secondary Outcome: Terminal Elimination Rate Constant (λz) of Vonoprazan
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/h
Arm/Group | Treatment A: Vonoprazan 20 mg Sprinkle Capsule on Pudding | Treatment B: Vonoprazan 20 mg Sprinkle Capsule on Applesauce | Treatment C: Vonoprazan 20 mg Tablet
Number analyzed (Participants) | 26 | 26 | 27
1/h | 0.0924 (19.5) | 0.0963 (18.4) | 0.0951 (16.0)

ADVERSE EVENTS:
Time Frame: Day 1 to Day 31
Description: All-cause mortality, serious and non-serious adverse events were measured in the safety population, which included all participants who received at least 1 dose of study drug. Safety data are presented for each treatment received, as pre-specified.
Arm/Group | Treatment A: Vonoprazan 20 mg Sprinkle Capsule on Pudding | Treatment B: Vonoprazan 20 mg Sprinkle Capsule on Applesauce | Treatment C: Vonoprazan 20 mg Tablet
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/26 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/26 | 0/27
Other Adverse Events (participants affected / at risk) | 2/26 | 2/26 | 4/27
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A: Vonoprazan 20 mg Sprinkle Capsule on Pudding (N=26) | Treatment B: Vonoprazan 20 mg Sprinkle Capsule on Applesauce (N=26) | Treatment C: Vonoprazan 20 mg Tablet (N=27)
Headache (Nervous system disorders) | 0 | 2 | 0
Muscle contractions involuntary (Nervous system disorders) | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1
Oral mucosal roughening (Gastrointestinal disorders) | 0 | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0
SARS-CoV-2 test positive (Investigations) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal investigators (PIs) are not permitted to publish the data. Data may be considered for reporting at a scientific meeting or for publication in a scientific journal. In these cases, the sponsor will be responsible for these activities and will work with the PIs to determine how the manuscript is written and edited, the number and order of authors, the publication to which it will be submitted, and any other related issues. The sponsor has final approval authority over all such issues.

DOCUMENTS (2):
  • Study Protocol (2022-04-25): https://cdn.clinicaltrials.gov/large-docs/38/NCT05366738/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-14): https://cdn.clinicaltrials.gov/large-docs/38/NCT05366738/SAP_001.pdf